CLINICAL TRIAL: NCT07134296
Title: MRI-guided Rectal Cancer Preservation Program
Brief Title: Magnetic Resonance Imaging (MRI)-Guided Rectal Cancer Preservation Program
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024.173
Record Dates: First submitted 2025-08-12; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Rectal Cancer
Keywords: TNT; MRI-guided Irradiation; Rectal Preservation
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose Escalation Phase (Experimental): Dose Escalation MR-guided TNT
  Interventions: Radiation: MR-Guided Irradiation

INTERVENTIONS:
Radiation: MR-Guided Irradiation — MR-Guided Irradiation

SUMMARY:
The goal of this clinical trial is to learn if the use of MRI-guided irradiation increases the rates of rectal preservation

DETAILED DESCRIPTION:
HYPOTHESIS

The implementation of Magnetic Resonance Image Guided Radiotherapy (MRgRT) into a TNT Program renders improved TME-free rates due to the better visualization and online dose-adaptation of the Gross Tumor Volume (GTV).

Rationale In the radiation setting, MRI provides superior soft tissue contrast compared to standard onboard X-ray imaging improving inter- and intra- observer delineation variation. MRgRT offers the opportunity to adapt the plan at each fraction to the anatomical changes seen. This is especially important in rectal cancer where the rectum is subject to interfractional position changes, volume shrinkage and intrafractional shape and size variation due to the variability in rectal filling.

Primary Objectives

A. To achieve 3-year TME-free survival of 75% while keeping 3-year DFS rates of 75%.

B. To achieve a CTCAE v5 grade 2-3 proctitis of less than 10% and grade 2-3 rectal bleeding rate of <2% at 2 years.

C. To achieve a Wexner Continence score of at least 90% over baseline at 2 years.

Secondary Objectives

A. Determination of blood and urine biomarkers of treatment response and toxicity .

B. Determination of radiomics biomarkers of treatment response and toxicity . C. Determination of rectal functionality with the Wexner Continence Score.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 or older with primary Stage II (T3-4, N0) or Stage III (any T, N1-2) biopsy-proven rectal cancer
* No prior radiation therapy to the target areas;
* ECOG 0-2 with medical status not contraindicating treatment with radical intent including TNT and TME (if required) and with basal laboratory values as follows:

  * Absolute neutrophil count (ANC) ≥ 1,000 cells/mm3
  * Platelets ≥ 50,000 cells/mm3.
  * Hemoglobin ≥ 8.0 g/dl.
  * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) < 4 x upper limit of normal.
  * Total bilirubin < 2 x upper normal mg/dL.
  * Alkaline phosphatase < 4 x upper limit of normal.

Exclusion Criteria:

* Patient unable to undergo an MRI examination

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2030-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Total Mesorectal Excision (TME)-free survival | 5-years
  To achieve 3-year TME-free survival of 75% while keeping 3-year DFS rates of 75%.

SECONDARY OUTCOMES:
Proctitis/Rectal Bleeding | 5-years
  To achieve a CTCAE v5 grade 2-3 proctitis of less than 10% and grade 2-3 rectal bleeding rate of <2% at 2 years.
Fecal Continence | 5-years
  To achieve a Wexner Continence score of at least 90% over baseline at 2 years.

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Martínez-Monge, M.D., Principal Investigator — Clínica Universidad de Navarra; Luis Fuertes, M.D., Principal Investigator — Clínica Universidad de Navarra

IPD SHARING:
Plan to Share IPD: Yes
On request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 5-years
Access Criteria: On request